CLINICAL TRIAL: NCT04210167
Title: Web-based Training and Telephone Follow-up of Patients With Heart Failure: Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Emine İLASLAN, lecturer, Akdeniz University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Akdeniz University 07
Record Dates: First submitted 2019-12-19; First posted 2019-12-24 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Heart Failure; Patient; Quality of Life; Symptoms
Keywords: heart failure; web-based training; telephone monitoring; symptom assessment; quality of life
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Intervention Model Description: This study is a randomized controlled study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- web-based training and telephone monitoring (Experimental): The heart failure patients in the intervention group were given web-based training for three months after discharge and followed up by telephone at the first, fourth, eighth and 12th weeks. At the same time, a text message was sent once a week. Scale data were collected before the patient was discharged from the hospital and at the third month of discharge.
  Interventions: Behavioral: web-based training and telephone monitoring

INTERVENTIONS:
Behavioral: web-based training and telephone monitoring — web-based training and telephone monitoring and short message

SUMMARY:
Web-based training and telephone monitoring have an effect on reducing symptom burden in patients with heart failure.

Web-based training and telephone monitoring have an effect on improving the quality of life of patients with heart failure.

Web-based training and telephone follow-up have an effect on reducing recurrent hospitalizations of patients with heart failure.

Web-based training and telephone follow-up have a positive effect on the clinical parameters (weight, waist circumference, blood pressure, creatinine) of patients with heart failure.

DETAILED DESCRIPTION:
The aim of this study was to determine the effect of web-based training and telephone monitoring on symptom management and quality of life in patients with heart failure. Study was conducted with the participation of 32 intervention and 32 control patients who have heart failure, in Akdeniz University Hospital Cardiology Clinic, between April 2018 and July 2019. Data were collected using the Patient Information Form, Left Ventricular Dysfunction Scale and Memorial Symptom Rating Scale-Heart Failure Scale, Website Analysis and Measurement Inventory. The patients in the intervention group received web-based training after discharge, and were followed up by telephone at the first, fourth, eighth and 12 weeks. The scale data were collected before the patient was discharged from hospital and at the third month of discharge.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing treatment at the Cardiology Clinic of Akdeniz University Hospital with a diagnosis of heart failure.
* Class I, II, III according to NYHA classification
* Has internet access and can use a computer / tablet or smartphone
* Agree to participate in the research

Exclusion Criteria:

* Functional class IV according to NYHA classification
* Diagnosed with psychiatric illness
* Malignancy diagnosed
* Visually and hearing impaired
* Diagnosed with chronic obstructive pulmonary disease

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
Has an effect on reducing symptom burden | 3 months
  Memorial Symptom Assessment Scale-Heart Failure: The Memorial Symptom Assessment Scale-Heart Failure was used to evaluate symptom prevalence, severity, and distress. For each of the 32 items, the patient indicated whether he/she had experienced the symptom by selecting "yes" or "no." If "yes" was selected, the severity of a symptom over the past 7 days was assessed using the response. The score range of each symptom is 0-4. Higher score indicates a higher symptom burden. Turkish version of the questionnaire was used.
Has an effect on improving quality of life | 3 months
  Left Ventricular Dysfunction Questionnaire: The questionnaire is a 36 item questionnaire for patients with left ventricular dysfunction. Responses are dichotomous (true or false). True responses are summed and the sum is expressed as a percentage. The score range of scale is 0-100. A higher score indicates a worse quality of life. Turkish version of the questionnaire was used.
Reducing heart failure patient rehospitalizations | 3 months
  Evaluation form of rehospitalizations: During the 3-month follow-up period, the number of admissions to the hospital and emergency outpatient clinic was recorded. In addition, if he was hospitalized, how many days he was hospitalized was recorded.
Positive effects on waist circumference | 3 months
  Waist circumference assessment form: The form was prepared by the researcher to record the waist circumference of the patients as "centimeters" unit.
Positive effects on weight | 3 months
  Weight assessment form: The form was prepared by the researcher to record the patients' weights in "kilogram" units.
Positive effects on blood pressure | 3 months
  Blood pressure assessment form: The form was prepared by the researcher to record the blood pressure of the patients as "mmHg" units
Positive effects on creatinine | 3 months
  Creatinine assessment form: A form was prepared by the researcher to record normal creatinine levels in the blood as "milligram" units.

CONTACTS AND LOCATIONS:
Overall Officials: Zeynep ÖZER, PhD, RN, Study Director — Akdeniz University
Locations (1):
- Akdeniz University, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD will share
Supporting Information: Study Protocol, SAP, CSR
Time Frame: starting 1 months after publication
Access Criteria: all people access

REFERENCES:
- [Background] Piamjariyakul U, Werkowitch M, Wick J, Russell C, Vacek JL, Smith CE. Caregiver coaching program effect: Reducing heart failure patient rehospitalizations and improving caregiver outcomes among African Americans. Heart Lung. 2015 Nov-Dec;44(6):466-73. doi: 10.1016/j.hrtlng.2015.07.007. Epub 2015 Aug 22. PMID 26307539
- [Background] Ponikowski P, Voors AA, Anker SD, Bueno H, Cleland JGF, Coats AJS, Falk V, Gonzalez-Juanatey JR, Harjola VP, Jankowska EA, Jessup M, Linde C, Nihoyannopoulos P, Parissis JT, Pieske B, Riley JP, Rosano GMC, Ruilope LM, Ruschitzka F, Rutten FH, van der Meer P. 2016 ESC Guidelines for the Diagnosis and Treatment of Acute and Chronic Heart Failure. Rev Esp Cardiol (Engl Ed). 2016 Dec;69(12):1167. doi: 10.1016/j.rec.2016.11.005. No abstract available. English, Spanish. PMID 27894487
- [Background] Seferovic PM, Stoerk S, Filippatos G, Mareev V, Kavoliuniene A, Ristic AD, Ponikowski P, McMurray J, Maggioni A, Ruschitzka F, van Veldhuisen DJ, Coats A, Piepoli M, McDonagh T, Riley J, Hoes A, Pieske B, Dobric M, Papp Z, Mebazaa A, Parissis J, Ben Gal T, Vinereanu D, Brito D, Altenberger J, Gatzov P, Milinkovic I, Hradec J, Trochu JN, Amir O, Moura B, Lainscak M, Comin J, Wikstrom G, Anker S; Committee of National Heart Failure Societies or Working Groups of the Heart Failure Association of the European Society of Cardiology. Organization of heart failure management in European Society of Cardiology member countries: survey of the Heart Failure Association of the European Society of Cardiology in collaboration with the Heart Failure National Societies/Working Groups. Eur J Heart Fail. 2013 Sep;15(9):947-59. doi: 10.1093/eurjhf/hft092. Epub 2013 Jun 19. PMID 23787723
- [Background] Wakefield B, Pham K, Scherubel M. Usability Evaluation of a Web-Based Symptom Monitoring Application for Heart Failure. West J Nurs Res. 2015 Jul;37(7):922-34. doi: 10.1177/0193945914568813. Epub 2015 Jan 26. PMID 25628261
- [Background] Wakefield BJ, Alexander G, Dohrmann M, Richardson J. Design and Evaluation of a Web-Based Symptom Monitoring Tool for Heart Failure. Comput Inform Nurs. 2017 May;35(5):248-254. doi: 10.1097/CIN.0000000000000324. PMID 28045703
- [Background] Yancy CW, Jessup M, Bozkurt B, Butler J, Casey DE Jr, Colvin MM, Drazner MH, Filippatos GS, Fonarow GC, Givertz MM, Hollenberg SM, Lindenfeld J, Masoudi FA, McBride PE, Peterson PN, Stevenson LW, Westlake C. 2017 ACC/AHA/HFSA Focused Update of the 2013 ACCF/AHA Guideline for the Management of Heart Failure: A Report of the American College of Cardiology/American Heart Association Task Force on Clinical Practice Guidelines and the Heart Failure Society of America. J Card Fail. 2017 Aug;23(8):628-651. doi: 10.1016/j.cardfail.2017.04.014. Epub 2017 Apr 28. No abstract available. PMID 28461259
- [Background] Zambroski CH, Moser DK, Bhat G, Ziegler C. Impact of symptom prevalence and symptom burden on quality of life in patients with heart failure. Eur J Cardiovasc Nurs. 2005 Sep;4(3):198-206. doi: 10.1016/j.ejcnurse.2005.03.010. PMID 15916924
- See also: American Heart Association, Warning Signs of Heart Failure — http://www.heart.org/HEARTORG/Conditions/HeartFailure/WarningSignsforHeartFailure/W